CLINICAL TRIAL: NCT03360604
Title: Utilizing Glycaemic Index: An Investigation of the Glycaemic Profiles and Cognitive Performance Displayed by Type 2 Diabetics Across the Course of a Day in Low and High Glycaemic Conditions
Brief Title: Utilizing Glycaemic Index: An Investigation of the Glycaemia and Cognition in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Grout (Other)
Responsible Party: Sponsor-Investigator, Matthew Grout, Doctoral Researcher, University of Reading
Organization: University of Reading (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017-151-DL
Record Dates: First submitted 2017-11-08; First posted 2017-12-04 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus, Type 2; Cognitive Impairment
Keywords: glycaemic index; glycaemia; diabetes mellitus; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: All participants took part in both conditions
Who Masked: Participant
Masking Description: Participants are not told which condition they are taking part in during each test day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low GI diet (Experimental): This diet consists of three meals (breakfast, lunch, snack) which all have a low glycaemic index. This is the Low Glycaemic Diet intervention.
  Interventions: Dietary Supplement: Low Glycaemic Diet
- High GI diet (Experimental): This diet consists of three meals (breakfast, lunch, snack) which all have a high glycaemic index. This is the High Glycaemic Diet intervention.
  Interventions: Dietary Supplement: High Glycaemic Diet

INTERVENTIONS:
Dietary Supplement: Low Glycaemic Diet — This intervention is a diet consisting of a Low GI breakfast, lunch and snack meal.
  Arms: Low GI diet
Dietary Supplement: High Glycaemic Diet — This intervention is a diet consisting of a High GI breakfast, lunch and snack meal.
  Arms: High GI diet

SUMMARY:
The current study aims to investigate the effects of two GI diets (low vs. high GI) in a sample (25 participants) that has diet controlled type 2 diabetes. This sample has been chosen as those with diabetes have been shown to suffer with poor glucose tolerance, along with the associated deficits such as compromised cognitive function. Therefore, it is expected that differences produced by the two diets on blood glucose concentrations and cognitive performance will be greater than those previously seen. If this is the case after analyzing the results, it will provide a potential strategy (diet) for improving glucose tolerance and cognitive performance in a vulnerable section of the population.

DETAILED DESCRIPTION:
With the introduction of the glycemic index in 1981, which can be defined as a measure of carbohydrate quality within foods, there has been a wealth of research into its' application to cognitive function. This research has been based on the theory that the availability of blood-borne glucose can have an impact on cognitive performance. This is supported by work that has shown that the brain consumes an immense amount of energy relative to the rest of the body, but possesses minute stores of glycogen which it could convert into its main energy source; glucose. This means the brain is reliant on the glucose supplied to it by the blood, which in turn requires the consumption of foods that can be broken down into glucose.

With this in mind, the vast majority of literature has focussed on the acute effects that foods differing in glycemic values may have on cognitive function, and have found many relevant findings such as less cognitive performance decline across the morning for children who eat a low GI breakfast. This could be explained as a low GI breakfast will contain higher quality carbohydrates, or in other words; slower absorbing carbohydrates, which would suggest the brain has access to a steady supply of glucose across the more.

Interesting work in the field of physiology has proposed the presence of a second meal effect, which can be defined as the glycemic index of a meal having an effect on the glycemic response to a subsequent meal. Surprisingly, there are very few pieces of psychology literature that investigate the possibility of a second cognitive meal effect, which is based on the theory that if a meals' GI can affect the glycemic response to a subsequent meal, then it may also have an effect on cognitive function. However, research into this has found some evidence for such an effect.

Although, there has been a wealth of research into the glycemic index as a whole, the methodology varies greatly from study to study. These problems are most evident when looking at the times that cognitive function tests are administered. For research based upon a theory that relies on availability of blood-borne glucose, the times of cognitive testing do not always align themselves with the time points that the glycemic response indicates are ideal testing times.

An initial study by the investigators looked to resolve the current lack of consistency amongst previous research by providing participants with three meals throughout the course of a day, whilst measuring blood glucose via finger prick. The aim was to identify where the biggest differences in blood glucose occur when looking at the results of a sample of 24 healthy participants. The time points identified would then provide information as to when significant differences in cognitive performance throughout the day may be expected.

A second study fed a larger healthy sample (40 participants) the same meals, but also included a cognitive task battery. Results from the blood glucose concentrations supported results from study 1, with the two diets producing measureable differences in the glycaemic profiles produced across a test day. This is another step into potentially producing a diet that could promote healthy glucose regulation and cognitive function.

The current study aims to investigate the effects of two GI diets (low vs. high GI) in a sample (25 participants) that has diet controlled type 2 diabetes. This sample has been chosen as those with diabetes have been shown to suffer with poor glucose tolerance, along with the associated deficits such as compromised cognitive function. Therefore, it is expected that differences produced by the two diets on blood glucose concentrations and cognitive performance will be greater than those previously seen. If this is the case after analyzing the results, it will provide a potential strategy (diet) for improving glucose tolerance and cognitive performance in a vulnerable section of the population.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 and 70 years of age.
* Willing to participate in the entire study.
* Male of female (not pregnant).
* Currently have type 2 diabetes mellitus.

Exclusion Criteria:

* Presence of any food intolerances or allergies.
* Being an elite athlete (very intense exercise more than 3 times a week).
* A history of drug or alcohol abuse.
* Presence of cancer.
* Presence of clinically diagnosed depression.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Change in cognitive performance on a Choice Reaction Time task | This test lasts 3 minutes. Participants are tested 9 times on each test day. There are two test days. Giving a total of 18 times, or approximately 54 minutes of performing this task across the entire study.
  Specifically, the number of errors and the reaction times of participants are recorded by the software that runs this task (E prime) as it is performed. The number of errors and the mean reaction times are later statistically assessed in SPSS.
Change in cognitive performance on a Rapid Visual Information Processing task | This test lasts 3 minutes. Participants are tested 9 times on each test day. There are two test days. Giving a total of 18 times, or approximately 54 minutes of performing this task across the entire study.
  Specifically, the number of errors and the reaction times of participants are recorded by the software that runs this task (E prime) as it is performed. The number of errors and the mean reaction times are later statistically assessed in SPSS.
Change in cognitive performance on a combined Choice Reaction Time and Rapid Visual Information Processing task | This test lasts 5 minutes. Participants are tested 9 times on each test day. There are two test days. Giving a total of 18 times, or approximately 90 minutes of performing this task across the entire study.
  Specifically, the number of errors and the reaction times of participants are recorded by the software that runs this task (E prime) as it is performed. The number of errors and the mean reaction times are later statistically assessed in SPSS.
Change in cognitive performance on a Letter Memory Task | This test lasts 5 minutes. Participants are tested 9 times on each test day. There are two test days. Giving a total of 18 times, or approximately 90 minutes of performing this task across the entire study.
  Specifically, the number of errors and the reaction times of participants are recorded by the software that runs this task (E prime) as it is performed. The number of errors and the mean reaction times are later statistically assessed in SPSS.

SECONDARY OUTCOMES:
Glycaemic profile | This is measured continuously throughout each day. Each day last approximately 9 hours. There are two test days. Giving a total of 18 hours of continuous glucose monitoring per participant.
  This is a participants' glucose concentration levels throughout the day, measured via a continuous glucose monitoring system.
Mood (alertness, anxiety and contentment) measured by Bond & Lader (1974) Visual Analogue Scale | This was measured 6 times a day (every 90 minutes starting at 0 minutes/baseline), giving a total of 12 times. Each time lasts approximately 5 minutes, giving a total of 60 minutes overall. Data will be reported for the duration of this 3 year PhD award.
  The Bond & Lader VAS provides participants with 16 lines measuring 100mm each. At the ends of each line are two words opposite in meaning. For example, 'alert' and 'drowsy'. A participant marks on the line closer to the word they currently feel. The score from each line is out of 0 to 100.
Sleepiness | This takes approximately 30 seconds to complete. Participants were tested six times a day. There were two test days. Giving a total of 12 times, or approximately 6 minutes overall.
  This was measured on a custom Visual Analogue Scale. Participants were presented with a 100mm line. At one end the word 'sleepy' appeared, and at the other end 'not sleepy' was present. Participants indicated how sleepy they felt by marking the line closer to the word they currently felt. Scores fell between 0 and 100.
Hunger | This takes approximately 30 seconds to complete. Participants were tested six times a day. There were two test days. Giving a total of 12 times, or approximately 6 minutes overall.
  This was measured on a custom Visual Analogue Scale. Participants were presented with a 100mm line. At one end the word 'hungry' appeared, and at the other end 'not hungry' was present. Participants indicated how hungry they felt by marking the line closer to the word they currently felt. Scores fell between 0 and 100.
Fullness | This takes approximately 30 seconds to complete. Participants were tested six times a day. There were two test days. Giving a total of 12 times, or approximately 6 minutes overall.
  This was measured on a custom Visual Analogue Scale. Participants were presented with a 100mm line. At one end the word 'full' appeared, and at the other end 'not full' was present. Participants indicated how full they felt by marking the line closer to the word they currently felt. Scores fell between 0 and 100.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Lamport, PhD, Principal Investigator — University of Reading; Matthew J Grout, PhD, Study Director — University of Reading; Julie A Lovegrove, PhD, Study Chair — University of Reading
Locations (1):
- Hugh Sinclair Unit, University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jenkins DJ, Wolever TM, Taylor RH, Barker H, Fielden H, Baldwin JM, Bowling AC, Newman HC, Jenkins AL, Goff DV. Glycemic index of foods: a physiological basis for carbohydrate exchange. Am J Clin Nutr. 1981 Mar;34(3):362-6. doi: 10.1093/ajcn/34.3.362. PMID 6259925
- [Background] Amiel SA. Nutrition of the brain: macronutrient supply. Proc Nutr Soc. 1994 Jul;53(2):401-5. doi: 10.1079/pns19940045. No abstract available. PMID 7972154
- [Background] Gomez-Pinilla F. Brain foods: the effects of nutrients on brain function. Nat Rev Neurosci. 2008 Jul;9(7):568-78. doi: 10.1038/nrn2421. PMID 18568016
- [Background] Ingwersen J, Defeyter MA, Kennedy DO, Wesnes KA, Scholey AB. A low glycaemic index breakfast cereal preferentially prevents children's cognitive performance from declining throughout the morning. Appetite. 2007 Jul;49(1):240-4. doi: 10.1016/j.appet.2006.06.009. Epub 2007 Jan 16. PMID 17224202
- [Background] Wolever TM, Jenkins DJ, Ocana AM, Rao VA, Collier GR. Second-meal effect: low-glycemic-index foods eaten at dinner improve subsequent breakfast glycemic response. Am J Clin Nutr. 1988 Oct;48(4):1041-7. doi: 10.1093/ajcn/48.4.1041. PMID 2844076
- [Background] Lamport DJ, Hoyle E, Lawton CL, Mansfield MW, Dye L. Evidence for a second meal cognitive effect: glycaemic responses to high and low glycaemic index evening meals are associated with cognition the following morning. Nutr Neurosci. 2011 Mar;14(2):66-71. doi: 10.1179/1476830511Y.0000000002. PMID 21605502
- [Background] Lamport DJ, Lawton CL, Mansfield MW, Moulin CA, Dye L. Type 2 diabetes and impaired glucose tolerance are associated with word memory source monitoring recollection deficits but not simple recognition familiarity deficits following water, low glycaemic load, and high glycaemic load breakfasts. Physiol Behav. 2014 Jan 30;124:54-60. doi: 10.1016/j.physbeh.2013.10.033. Epub 2013 Oct 30. PMID 24184411
- [Derived] Grout M, Lovegrove JA, Lamport DJ. A multimeal paradigm producing a low glycemic response is associated with modest cognitive benefits relative to a high glycemic response: a randomized, crossover trial in patients with type 2 diabetes. Am J Clin Nutr. 2023 May;117(5):859-869. doi: 10.1016/j.ajcnut.2023.02.017. Epub 2023 Feb 24. PMID 36841444